CLINICAL TRIAL: NCT02135289
Title: The Role of Interferon Gamma Releasing Assays (IGRA) in Screening and Monitoring for Tuberculosis During Anti-TNF Therapy in Patients With Immune-mediated Inflammatory Disease (IMID)
Brief Title: The Role of IGRA in Screening and Monitoring for TB During Anti TNF Therapy in Patients With IMID
Acronym: IGRA
Status: Completed | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Siew Chien NG, Professor, Chinese University of Hong Kong
Other Study IDs: IGRA
Record Dates: First submitted 2014-04-29; First posted 2014-05-09 (Estimated); Last update posted 2020-04-29 (Actual); Status verified 2020-04

CONDITIONS: Inflammatory Bowel Disease; Crohn Disease; Ulcerative Colitis; Tuberculosis; Immune-mediated Inflammatory Disease
MeSH Terms: conditions — Inflammatory Bowel Diseases; Crohn Disease; Colitis, Ulcerative; Tuberculosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- IMID patients: Patients with IMID
- Control - subjects without IBD: Patients without IBD

SUMMARY:
Hong Kong is a region of intermediate TB burden, and the reactivation of latent TB in IMID patients treated with anti-TNF can be a serious problem. This study aims to investigate the role of IGRA in screening for latent TB in IBD patients and control subjects. In part II of the study, patients of other immune-mediated inflammatory diseases (IMID) will also be included to investigate the role of serial interferon-gamma release assays (IGRA) for the diagnosis of tuberculosis (TB) infection in patients with immune-mediated inflammatory diseases (IMID) treated with biologics

DETAILED DESCRIPTION:
The incidence of inflammatory bowel disease is rising in Hong Kong. Anti-tumor necrosis factor alpha (anti-TNF)-α is effective and increasingly being used for the treatment of patients with refractory disease and complicated disease behaviour. The reactivation of latent tuberculosis (TB) is a well-recognised complication associated with the use of anti-TNF therapy, and most cases occurred in endemic regions. Hong Kong is a region of intermediate TB burden, and the reactivation of latent TB in IMID patients treated with anti-TNF can be a serious problem. Screening has been shown to reduce the incidence of TB, but it remains unclear whether monitoring during anti-TNF therapy is effective. Despite reported efficacy with the current screening strategy, active TB developed in up to 11.4% of patients receiving anti-TNF therapy. There is therefore an urgent need for better disease monitoring and prevention, particularly in regions where TB is endemic.

Part I of this study aims to investigate the role of IGRA in screening for latent TB in IBD patients and control subjects. Part II of this study is a prospective study of serial interferon-gamma release assays (IGRA) for the diagnosis of tuberculosis (TB) infection in patients with immune-mediated inflammatory diseases (IMID) treated with biologics

ELIGIBILITY:
Inclusion Criteria:

* patients aged 18 years or older
* patients with a diagnosis of Crohn's disease (CD) or ulcerative colitis (UC) for at least 3 months defined by histology or radiology

Exclusion Criteria:

* Patients with a previous history of TB
* Patients with a positive IGRA or CXR suggesting latent tuberculosis prior to commencement of therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients attending Prince of Wales Hospital
Sampling Method: Non-Probability Sample
Enrollment: 9160 (Actual)
Dates: Start 2012-03 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
IGRA positivity | 2 Years
  The comparison of IGRA positivity between treatment-naïve IBD patients, IBD patients on immunosuppressive drugs, and healthy controls
IGRA conversion | 3 Years
  The proportion and outcome of patients with IGRA conversion during anti-TNF therapy or receiving other immunosuppressive drugs

CONTACTS AND LOCATIONS:
Overall Officials: Siew Chien Ng, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No